CLINICAL TRIAL: NCT05395923
Title: The Effects of Palatal Pre-sutures on Hemostasis and Patient Comfort in Connective Tıssue Graft Surgery
Brief Title: The Effects of Palatal Pre-sutures in Connective Tıssue Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Principal Investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-KAEK-58-22-01
Record Dates: First submitted 2022-04-03; First posted 2022-05-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Suture, Complication; Gingival Recession; Bleeding Hemorrhage
MeSH Terms: conditions — Gingival Recession; Hemorrhage | interventions — Sutures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palatal Pre-Suture (GPCS) (Experimental): In the test group, GPCS (Silk, 4-0, 18 mm, 3/8 sharp needle) will be placed before the incision in the palatal region. GPCS will be taken one week after surgery.
  Interventions: Procedure: Suture
- No Palatal Suture (No GPCS) - Control (Active Comparator): In the control group, no sutures will be applied before graft harvesting from the palate.
  Interventions: Procedure: No Suture CTG -Control

INTERVENTIONS:
Procedure: Suture — The pressure application will be applied before the incision on the palate.
  Arms: Palatal Pre-Suture (GPCS)
Procedure: No Suture CTG -Control — A graft will be taken from the palate before the procedure is applied.
  Arms: No Palatal Suture (No GPCS) - Control

SUMMARY:
Connective tissue graft operation is one of the most frequently performed surgical procedures to increase the width of the attached gingiva and to treat gingival recessions. The most preferred donor site during this operation is the palatal mucosa.Reported postoperative complications are usually related to the donor site. Problems such as prolongation of bleeding time, delay in wound healing and severe pain in the palatal region where the graft is taken are frequently encountered. Bleeding control in the palatal donor area is very important for patient comfort. Additional measures may be required to control bleeding, such as sutures with or without hemostatic agents, or acrylic, plastic palatal stents and periodontal pastes prepared before the operation. Suturing the Greater Palatine Artery (GPA) or terminal vessel branches has been shown to be an effective method to control palatal bleeding.

Therefore the aim of this study is to evaluate the effectiveness of the pre-suture method applied in the palatal region before the connective tissue graft is taken in reducing hemostasis.Pre-suture method can increase the operator's field of vision and operational comfort. Patient-reported outcomes such as the amount of pain and bleeding in the palatal donor area during and after surgery, painkiller intake, number of days of discomfort, satisfaction, quality of life, and willingness to be treated will be evaluated.

In addition, it will be evaluated whether this suture technique affects the healing of the half-thickness flap in the palatal region after obtaining a connective tissue graft with a single incision method.

DETAILED DESCRIPTION:
Various methods have been described to manage bleeding and/or promote healing of the palatal donor site.These techniques include sutures with or without hemostatic agents, or the use of materials such as acrylic or plastic palatal stents, periodontal seals, and platelet-rich fibrin (PRF) prepared before the operation. The use of an additional hemostatic agent often requires additional surgical time and expense, and most of the techniques described in the literature for the management of palatal hemorrhage are used to control bleeding after it has occurred. GPA and/or suturing of terminal vessel branches is a popular and effective technique to control palatal bleeding.Recently, a detailed protocol for a Greater Palatine Compression Suture (GPCS) has been presented and proposed as a predictable method for controlling bleeding when this suture is applied preoperatively at the palatal donor site. This protocol is based on the estimated location of the greater palatal foramen and vascular bundle and has proven to be efficient in controlling palatal bleeding. The recommended protocol for GPCS is as follows:

1. The midpalatal line is defined.
2. An imaginary line is joined to the midpalatal line from the midline of the first and second maxillary molars (point X).
3. Another point (Point A) is defined along the X line at a distance of 20 mm from the midpalatal line. (Y point)
4. The needle is passed through point A along its curve, and the exit point (point B) of the needle should be approximately 10 mm medial and approximately 5 mm anterior to point A. 1/2 diameter, triangular body, 3-0 braided silk sutures recommended in this protocol were used. The effectiveness of GPCS on palatal hemostasis before obtaining a free gingival graft was also evaluated previously. Reduced palatal bleeding is a valuable clinical benefit in terms of reduced perioperative morbidity, better visibility for the operator, reduced need for hemostatic agents, and operation time.

In addition, the availability of such a technique can be reassuring to the operator when removing autogenous grafts and may be of additional importance in patients prone to bleeding. One of the primary results in our study was the amount of perioperative bleeding. Methods of measuring perioperative blood loss include direct volumetric estimation, weighing blood gauze pads, using various formulas based on hematocrit values, and visual estimation. In our study, bloody gauze pads will be measured with precision scales and the amount of bleeding in the palate will be directly measured during the operation.

In our study, it is aimed to evaluate whether the BPKS technique has any effect on the healing of the half-thickness flap in the donor area when applied in connective tissue graft procedures obtained with the single incision method.

Evaluation of donor site wound healing with anamnesis and index records will be performed by a blinded investigator who did not perform the operation (B.K.).

Initial periodontal treatments will be performed for each patient participating in the study before surgical procedures. Oral hygiene, scaling, root planing and occlusal adjustments will be carried out when necessary. Connective tissue graft will be harvested with a single incision method. Surgical procedures will be performed by a single investigator (M.Z.).

At the beginning of the operation, 0.5 mL of 2% lidocaine anesthesia containing 1:200,000 adrenaline will be administered to the palatal donor area to both the control and test groups, from the points corresponding to the canine and the first molar. In the test group, GPCS (Silk, 4-0, 18 mm, 3/8 sharp needle) will be placed before the incision in the palatal region. Then, connective tissue graft will be taken with a single incision technique using a 15-C scalpel in both groups. The thickness of the connective tissue graft to be taken in our study will be 1.5-2 mm, and its dimensions will be 8X8 mm as standard. Then, the half-thickness flap in the palatal region will be closed with a continuous locked suture (Trofilen, 5/0, 16 mm, 3/8 sharp needle). The connective tissue graft will be sutured to the recipient area with 6-0 polyglactin sutures (Pegalak rapid, 13 mm, 3/8 sharp needle) and the flap is shifted coronally (Trofilen, 5/0, 16 mm, 3/8 sharp needle) will be closed with. Measurement of blood loss will be carried out as described above.

There is no study that applies the BPKS technique during the connective tissue graft operation. In addition, patient-reported outcome measures such as painkiller intake, number of days of discomfort, satisfaction, quality of life, and willingness to be treated again, as well as the amount of pain and bleeding of the palatal donor site during and after surgery, were not examined.

The operation period will be started after the incision and will be terminated when the operation is completed. For postoperative care, the patient will be prescribed a mouthwash containing 0.12% chlorhexidine digluconate to be used twice a day for 3 weeks. In addition, analgesic (Flurbiprofen 100 mg film tablet) will be prescribed to be used when they feel pain. After the operation, patients will be asked not to brush the operation area for 2 weeks and patients will be warned to avoid hard chewing. Brushing with a soft brush will be required in the 3rd postoperative week. The suture in the donor area will be removed in the 1st week, and the suture in the recipient area will be removed in the 2nd week postoperatively. GPCS will be taken 1 week after the operation.

Patients will be called for controls on the 3rd day, 1st and 2nd weeks, 1st, 3rd and 6th months after the operation and their measurements will be recorded. The scales evaluated by the patient will be given to the patient after the operation and will be collected when the study is finished. The records that the physician should take after the surgery will always be recorded by a single researcher. The investigator who took the records will not know the surgical technique applied.

ELIGIBILITY:
Inclusion Criteria:

* - The patient must be over the age of 18,
* Not having any systemic disease,
* Not receiving chemotherapy or radiotherapy treatment,
* Not using drugs regularly and not being addicted to drugs,
* Not be in pregnancy and/or lactation period,
* Not smoking,
* Not having received antibiotic treatment in the last 6 months,
* Presence of Cairo Type 1 or Type 2 recession defect in a single tooth,
* The patient is cooperative.

Exclusion Criteria:

* The patient is younger than 18 years old,
* Active infectious disease (acute hepatitis, AIDS, tuberculosis), cancer or any systemic condition that may affect periodontal tissues,
* Receiving chemotherapy or radiotherapy treatment,
* Being on regular medication and being addicted to drugs,
* Patients with a plaque score greater than 20% after phase I treatment (Silness and Löe, 1964),
* Being in pregnancy and/or lactation period,
* Being a smoker
* To have been treated with antibiotics in the last 6 months,
* Not being cooperative.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Measuring the Amount of Intra-operative Bleeding with a Precision Balance | During surgery
  In our study, the amount of blood lost will be estimated by using the gauze weight method, which is a method of directly estimating blood loss. All measurements will be made on a 1 g precision digital balance. Sterile gauze swabs will be weighed dry before the operation. The gauze pads that will be used later will be moistened with 10 mL of sterile 0.9 g/L saline solution before starting the procedure and the weight will be measured again. The time from the removal of the connective tissue graft to the end of the operation will be measured and the pre-moistened gauze pads will be used on the palate during this period and will be stored separately and their weight will be measured immediately after the operation is over. In this method, aspiration in the palatal region should be avoided to minimize errors in blood loss measurement.
Reporting of secondary bleeding as present/absent in the 1st postoperative week | 1st postoperative week after the operation.
  Reporting of secondary bleeding as present/absent both by the patient and by the physician in the follow-up appointments in the 1st postoperative weeks
patient discomfort and satisfaction [Oral Health Impact Profile ] | On the 3rd day after the operation.
  In this evaluation, the Oral Health Impact Profile (OHIP-14) test will be used by marking the patients on the 3rd postoperative day.
  Likert response system in the evaluation of the OHIP14 scale:
  0: "never",
  1. "very little"
  2. "sometimes"
  3. "quite often"
  4. is rated as "often". The total score of the answers given by the participant to each item is evaluated by calculating.
  The total score is minimum 0, maximum 56. It is concluded that as the total score increases, the severity of the problem increases and the quality of life decreases.
Evaluation of the pain felt by the patients after the operation with Visual Analogue Scale | 3rd day after the operation.
  Pain scores will be recorded on the postoperative 3rd day. It is determined by the patient's assessment of the intensity of pain felt on a scale from 0 to 10.
  0: No pain, 10: There is unbearable pain.
Reporting of secondary bleeding as present/absent in the 2nd postoperative week | 2nd postoperative week after the operation.
  Reporting of secondary bleeding as present/absent both by the patient and by the physician in the follow-up appointments in the 2nd postoperative weeks
patient discomfort and satisfaction [Oral Health Impact Profile ] | 1st week after the operation.
  In this evaluation, the Oral Health Impact Profile (OHIP-14) test will be used by marking the patients on the 1st postoperative week.
  Likert response system in the evaluation of the OHIP14 scale:
  0: "never",
  1. "very little"
  2. "sometimes"
  3. "quite often"
  4. is rated as "often". The total score of the answers given by the participant to each item is evaluated by calculating.
  The total score is minimum 0, maximum 56. It is concluded that as the total score increases, the severity of the problem increases and the quality of life decreases.
patient discomfort and satisfaction [Oral Health Impact Profile ] | 2nd week after the operation.
  In this evaluation, the Oral Health Impact Profile (OHIP-14) test will be used by marking the patients on the 2nd postoperative week.
  Likert response system in the evaluation of the OHIP14 scale:
  0: "never",
  1. "very little"
  2. "sometimes"
  3. "quite often"
  4. is rated as "often". The total score of the answers given by the participant to each item is evaluated by calculating.
  The total score is minimum 0, maximum 56. It is concluded that as the total score increases, the severity of the problem increases and the quality of life decreases.
patient discomfort and satisfaction [Oral Health Impact Profile ] | 4th week after the operation.
  In this evaluation, the Oral Health Impact Profile (OHIP-14) test will be used by marking the patients on the 4th postoperative week.
  Likert response system in the evaluation of the OHIP14 scale:
  0: "never",
  1. "very little"
  2. "sometimes"
  3. "quite often"
  4. is rated as "often". The total score of the answers given by the participant to each item is evaluated by calculating.
  The total score is minimum 0, maximum 56. It is concluded that as the total score increases, the severity of the problem increases and the quality of life decreases.
Evaluation of the pain felt by the patients after the operation with Visual Analogue Scale | 1st week after the operation.
  Pain scores will be recorded on the postoperative 1st week by marking the Visual Analogue Scale (VAS). It will be determined on a scale from 0 (no pain) to 10 (unbearable pain).
  It is determined by the patient's assessment of the intensity of pain felt on a scale from 0 to 10.
  0: No pain 10: There is unbearable pain
Evaluation of the pain felt by the patients after the operation with Visual Analogue Scale. | 2nd week after the operation.
  Pain scores will be recorded on the postoperative 2nd week by marking the Visual Analogue Scale (VAS). It will be determined on a scale from 0 (no pain) to 10 (unbearable pain).
  It is determined by the patient's assessment of the intensity of pain felt on a scale from 0 to 10.
  0: No pain, 10: There is unbearable pain.
Evaluation of the pain felt by the patients after the operation with Visual Analogue Scale | 4th week after the operation.
  Pain scores will be recorded on the postoperative 4th week by marking the Visual Analogue Scale (VAS). It will be determined on a scale from 0 (no pain) to 10 (unbearable pain).
  It is determined by the patient's assessment of the intensity of pain felt on a scale from 0 to 10.
  0: No pain, 10: There is unbearable pain.

SECONDARY OUTCOMES:
Evaluation of palatal wound healing by measuring the Early Wound Healing Index in the first 3 months after the operation | 3rd day after surgery.
  Early Wound Healing Score (EHS): After the operation, the wound area will be evaluated with EHS on the 3rd day. The EWHS consists of three parameters:
  A) Clinical signs of re-epithelialization: -Converged incision edges: 6 points, - Contact incision edges: 3 points, - Visible distance between incision edges: will be evaluated as 0 points.
  B) Clinical signs of hemostasis: - Absence of fibrin at the incision margins: 2 points, - Presence of fibrin at the incision margins: 1 point, - Bleeding at incision margins: 0 points C) Clinical signs of inflammation: - Absence of redness throughout the incision: 2 points, - Redness involving <50% of the incision length: 1 point, - Redness and/or significant swelling involving >50% of the incision length: 0 points. For ideal wound healing, all scores in A, B, and C are added together and the highest score of 10 is considered as the best healing, and the score of 0 for the worst wound healing.
Findings of necrosis on the donor area | During and first 3 months after surgery
  Evaluation by the patient by conducting a survey as yes/no
Findings of healing with complications on the donor area | During and first 3 months after surgery
  Evaluation by the patient by conducting a survey as yes/no
Evaluation of palatal wound healing by measuring the Early Wound Healing Index | 1st week after surgery.
  Early Wound Healing Score (EHS) :After the operation, the wound area will be evaluated with EHS on the 1st week after surgery. The EHS consists of three parameters:
  A) Clinical signs of re-epithelialization: -Converged incision edges: 6 points, - Contact incision edges: 3 points, - Visible distance between incision edges: will be evaluated as 0 points.
  B) Clinical signs of hemostasis: - Absence of fibrin at the incision margins: 2 points, - Presence of fibrin at the incision margins: 1 point, - Bleeding at incision margins: 0 points C) Clinical signs of inflammation: - Absence of redness throughout the incision: 2 points, - Redness involving <50% of the incision length: 1 point, - Redness and/or significant swelling involving >50% of the incision length: 0 points. For ideal wound healing, all scores in A, B, and C are added together and the highest score of 10 is considered as the best healing, and the score of 0 for the worst wound healing.
Evaluation of palatal wound healing by measuring the Early Wound Healing Index | 2nd week after surgery.
  Early Wound Healing Score (EHS) :After the operation, the wound area will be evaluated with EHS on the 2nd week after surgery. The EHS consists of three parameters:
  A) Clinical signs of re-epithelialization: -Converged incision edges: 6 points, - Contact incision edges: 3 points, - Visible distance between incision edges: will be evaluated as 0 points.
  B) Clinical signs of hemostasis: - Absence of fibrin at the incision margins: 2 points, - Presence of fibrin at the incision margins: 1 point, - Bleeding at incision margins: 0 points C) Clinical signs of inflammation: - Absence of redness throughout the incision: 2 points, - Redness involving <50% of the incision length: 1 point, - Redness and/or significant swelling involving >50% of the incision length: 0 points. For ideal wound healing, all scores in A, B, and C are added together and the highest score of 10 is considered as the best healing, and the score of 0 for the worst wound healing.
Evaluation of palatal wound healing by measuring the Early Wound Healing Index | 1st month after surgery.
  Early Wound Healing Score (EHS) :After the operation, the wound area will be evaluated with EHS on the 1st month after surgery. The EHS consists of three parameters:
  A) Clinical signs of re-epithelialization: -Converged incision edges: 6 points, - Contact incision edges: 3 points, - Visible distance between incision edges: will be evaluated as 0 points.
  B) Clinical signs of hemostasis: - Absence of fibrin at the incision margins: 2 points, - Presence of fibrin at the incision margins: 1 point, - Bleeding at incision margins: 0 points C) Clinical signs of inflammation: - Absence of redness throughout the incision: 2 points, - Redness involving <50% of the incision length: 1 point, - Redness and/or significant swelling involving >50% of the incision length: 0 points. For ideal wound healing, all scores in A, B, and C are added together and the highest score of 10 is considered as the best healing, and the score of 0 for the worst wound healing.
Findings of necrosis on the donor area | During and first 3 months after surgery
  Evaluation by the physician by conducting a survey as yes/no
Findings of healing with complications on the donor area | During and first 3 months after surgery
  Evaluation by the physician by conducting a survey as yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Karaduman, Principal Investigator — bkaraduman@biruni.edu.tr
Locations (1):
- Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No